CLINICAL TRIAL: NCT02357927
Title: A Single Session Intervention For Fear Of Recurrence In Breast Cancer Patients (The Mini AFTERc): A Controlled Trial
Brief Title: A Single Session Intervention For Fear Of Recurrence In Breast Cancer Patients
Acronym: Mini-AFTER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of St Andrews (Other)
Responsible Party: Principal Investigator, Prof G Humphris, Chair of Health Psychology, University of St Andrews
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: StAMedSchoolSEC
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Fear
Keywords: fears of recurrence; cancer; brief intervention; telephone counseling; following primary cancer treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Placebo Comparator): simple general telephone call
  Interventions: Behavioral: telephone call
- Mini-AFTERc Intervention (Experimental): 20-30 minute structured conversation with breast cancer patient using Mini-AFTERc Manual
  Interventions: Behavioral: Mini-AFTERc

INTERVENTIONS:
Behavioral: Mini-AFTERc — 20-30 minute structured conversation following guidelines and instruction within the Mini-AFTERc 20 page manual
  Arms: Mini-AFTERc Intervention
Behavioral: telephone call — this consists of a 20-30 minute conversation about the general well-being of the patient with no specific reference to recurrence fears unless raised by the patient explicitly themselves
  Arms: control

SUMMARY:
This is a controlled trial of the Mini-AFTERc intervention to reduce fears of recurrence in breast cancer patients. The sample will be collected in NHS Fife Breast Cancer Services (n=32). The intervention is a short telephone counseling service of 20 minutes delivered by the patient's breast cancer specialist nurse. Dependent measures consist of the ACCRE FoR 4 item measure and the EORTC Intervention overall satisfaction scale.

DETAILED DESCRIPTION:
1. Background The majority of breast cancer patients completes successfully their treatment and therefore become survivors with some of them experience negative outcomes. One of the most prevalent unmet needs of the breast cancer survivors is Fear of Recurrence. Fear of Cancer Recurrence is defined as "the fear or worry that cancer will return, progress or metastasise". More specifically, 33% to 96% of the patients report FoR of cancer, while in 9% to 34% of these patients, the fear of recurrence is so detrimental even to their lives. Women of younger age with children have reported to have more severe FCR .

   Findings suggest that FoR can remain stable in cancer survivors five years or more after the diagnosis . Research has shown that cancer survivors that experience FoR, suffer from psychological and affective difficulties because of their initial worries of being cancer patients a second time. The most frequent of these negative outcomes are distress, stress-response symptoms and lower quality of life. Consequently, there is much interest of the researchers to focus on the factors that influence FoR in cancer patients, and the effect of FoR in survivors' quality of life . Less research has focused on interventions that can reduce fear of recurrence in cancer patients. The AFTER intervention is one of them, conducted a systematic intervention. The intervention was successful, since the study reported reduction in FoR at 6 month follow-up.

   The aim of the current study is to examine the effect of the Mini-AFTERc intervention, which is a shorter version of AFTER intervention, in reduction of fear of recurrence in breast cancer survivors with moderate level of FoR in comparison with a control group, where as the full AFTER intervention target patients with more severe FoR.
2. Research Question Whether the single-session intervention Mini AFTERc, delivered by a phone call, can reduce fear of recurrence in breast cancer patients with moderate level of fear in contrast with a control group.
3. Hypothesis The mini AFTERc intervention will reduce fear of recurrence in breast cancer patients with moderate level of fear, whereas FoR will not be reduced in the control group.
4. Methods and materials 4.1 Study design The study will be a quasi-experiment design implementing a single-session intervention which is aimed at reducing fear of recurrence in breast cancer patients with moderate level of fear, whereas FoR will not be reduced in the comparison group.

   4.2 Location of study The location of the study will be at NHS fife, Breast Cancer Unit of Queen Margaret Hospital, Dunfermline, where breast cancer patients can be treated and supported. Three experienced nurses of this unit will employ the Mini-AFTERc intervention.

   4.3 Participants Patients of NHS fife, Breast Cancer Unit of Queen Margaret Hospital, Dunfermline, in order to be included in the study, have to be breast cancer patients who have completed primary treatment and are worried about fear of cancer recurrence. An estimated number of participants are 34 patients to be able to answer successfully the research question. More specifically, the 17 patients of the treated group will receive a structured phone, based on the mini AFTERc intervention, whereas call the 17 patients of the control group will receive a standard phone call, which will not be a mini- After. A power analysis was conducted using NQueryAdvisor. A sample size of 17 in each group will have 80% power to detect a difference in means of 4 on the four item Fears of Recurrence Scale (the difference between the Control group mean: 25 and a Intervention group mean: 21) assuming that the common standard deviation is 4 using a two group t-test with a 0.05 two-sided significance level. Values obtained of SD and likely effect size from unpublished data held by Ozakinci and Humphris of breast and colorectal cancer patients and the original feasibility study conducted by Davidson and Humphris.

   All patients of the unit are welcome to participate. Participants will be invited in the study after the primary treatment, during a routine-care follow-up. The information sheet, the consent form and a pre-paid envelope will be provided in the patients. After they have completed the consent form, they will complete the questionnaire measure of FoR severity (ACCRE), in which they have to score above the cut-off to be included in the study.

   4.4 Measures and intervention The severity of FoR will be measured by employing the 4-item severity scale ACCRE at baseline and at 1-month follow-up. The second outcome measure will be the EORTC Satisfaction of Intervention measuring the overall satisfaction of the patients. The study will employ the Mini-AFTERc intervention, which is based on the six-session full AFTER intervention. The AFTER intervention was initially developed for head and neck patients to be targeted as patients with high level of FoR.

   The Mini-AFTERc intervention is a single-session, cognitive behavioral intervention based on the Leventhal's Self-Regulation Model and has been designed to be used with patients who report moderate levels of FoR. The aim of the intervention is to normalize and reduce FoR to a manageable level but still facilitate patients to be aware of the risks. The patients are enabled to be vigilant in symptoms change.
5. Data analysis The audio recording of the intervention consultation will be transcribed. Analysis of pre and post tests will be conducted by SPSS Predictive Analytics software v.21. The post-test will be subtracted from the pre-test to derive a change score. An analysis of variance will be conducted with a number of covariates (i.e. age and disease severity). The dependent variable will be the FoR ACCRE change score
6. Ethical approval

   The National Research Ethics Service will be contacted to prepare the NRES form and NHS Fife R&D Governance forms as the study will be conducted with NHS Fife.

   Furthermore, we need to apply UTREC Ethics for the University of St Andrews, too.
7. Governance of study and support of participants The research project will be supervised by Professor Gerry Humphris. If needed, additional support to the patients will be provided by The Psychological Services at Edinburgh Cancer Unit, where Professor Humphris is a honorary clinical psychology consultant to the service and can pick up these referrals.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patient completed treatment
* female

Exclusion Criteria:

* psychiatric illness
* cognitive deficit (e.g. dementia)
* no access to telephone

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
ACCRE 4-Item Fears of Recurrence Questionaire | 1 month

SECONDARY OUTCOMES:
EORTC Intervention satisfaction single global item | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Humphris, PhD, Principal Investigator — University of St Andrews
Locations (1):
- Breast Cancer Services, Queen Margaret Hospital, Dunfermline, Fife, United Kingdom

REFERENCES:
- [Background] Humphris G, Ozakinci G. The AFTER intervention: a structured psychological approach to reduce fears of recurrence in patients with head and neck cancer. Br J Health Psychol. 2008 May;13(Pt 2):223-30. doi: 10.1348/135910708X283751. PMID 18492319